CLINICAL TRIAL: NCT05172297
Title: A Non-randomized Controlled Trial of the Effects of an Internet-delivered Parent Training Intervention (Parent Web) at the Transition to Early Adolescence for Parents of Children That Have Participated in Preschool PATHS®
Brief Title: Internet-based Universal Parent Training as a Booster to PATHS®: Parent Web
Acronym: PW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Responsible Party: Principal Investigator, Laura Ferrer Wreder, Associate Professor of Psychology, Stockholm University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FoUI-940010
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Family Conflict; Family Relations; Family Dysfunction
Keywords: parent training; universal; youth externalizing problems; family conflict; warmth in families

STUDY DESIGN:
Intervention Model Description: This is a non-randomized controlled experiment (i.e., quasi-experiment) with a wait-list comparison group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Experimental): The immediate intervention group will take part in the online parent training program called the Parent Web (PW). This immediate intervention group are parents of PATHS children who took part in a social emotional curriculum (PATHS) at age 4 to 5 years old and during the PW trial will be 11 to 13 years old. Parents are participating in the Parent Web.
  Interventions: Behavioral: Parent Web
- Wait-List Control Group (Other): This is a group of parents who are in a wait-list control group and will receive the Parent Web, after pre and post testing.
  Interventions: Behavioral: Parent Web

INTERVENTIONS:
Behavioral: Parent Web — Parent-Web (PW) is internet delivered and rooted in social learning and coercion theory, PW supports parenting practices and parent-child interactions encouraging prosocial behavior and emotion regulation, reduce coercive parenting, improve communication, problem solving, and warmth. PW has a universal and selective edition. Universal PW has 5 basic modules (1 module per week, 6-8 weeks) and bonus modules. Basic modules contain information, exercises, and videos of actors showing parenting practices. A family guide supports parents through modules.

SUMMARY:
To test an online parent training program. Relative to a matched comparison, those in the Parent Web (PW) will show benefits on well-being, parenting, stress, youth mental health. Parents of PATHS children are the immediate intervention group.

DETAILED DESCRIPTION:
Parent-Web (PW) is internet delivered and rooted in social learning and coercion theory, PW supports parenting practices and parent-child interactions encouraging prosocial behavior and emotion regulation, reduce coercive parenting, improve communication, problem solving, and warmth. PW has a universal and selective edition. Universal PW has 5 basic modules (1 module per week, 6-8 weeks) and bonus modules. Basic modules contain information, exercises, and videos of actors showing parenting practices. A family guide supports PW participants through PW modules. No published outcome evaluations of universal PW currently exist. However, benefits were found for selective PW. This study will test the effects of universal PW as a booster to PATHS (Promoting Alternative Thinking Strategies) a universal school-based intervention designed to enhance child social emotional competence. All PW trial participants are parents to at least one adolescent child (aged 11-13). Immediate PW participants are parents who have a child that participated in PATHS at age 4-5 years old.

ELIGIBILITY:
Inclusion Criteria:

Immediate intervention group are parents of children aged 11-13 who participated in PATHS at age 4-5 years old.

Parents in the wait list comparison group have children who are matched to the children of parents in the immediate intervention group.

Matching criteria are:

Wait-list group parents' child's present-day gender (matching criteria 1) is the same as the matched child who's parents are in the immediate intervention group, wait-list group parents' child's present-day age is similar to the matched child who's parents are in the immediate intervention group, namely child birthdays within 6 months of each other (matching criteria 2), and wait-list group parents' children live in the same postal code as the matched immediate intervention group child (matching criteria 3), and matched children have all lived in Sweden since 2014 (matching criteria 4). If these 4-matching criteria are too restrictive and do not provide enough matches to recruit from, then the matching criteria will be reduced to points 1, 2, and point 3. Children do not participate in the Parent Web intervention trial, but parents of children do participate.

Exclusion Criteria: See inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Parents in the wait list comparison group have children who are matched to the children of parents in the immediate intervention group. And one of the matching criteria are: Wait-list group parents' child's present-day gender is the same as the matched child who's parents are in the immediate intervention group
Enrollment: 163 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in parent rating of child's emotional problems, conduct problems, hyperactivity, peer problems and prosocial behavior | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rating of their child's emotional problems, conduct problems, hyperactivity, peer problems and prosocial behavior as indexed by the Strengths and Difficulties Questionnaire (SDQ). The SDQ consists of 25 items rated on a 3-point Likert scale with response options that range from 0 = not true, 1 = somewhat true, 2 = certainly true. Higher scores indicate a worse outcome on the emotional problems, conduct problems, hyperactivity, peer problems scale scores. Higher scores on the prosocial behavior scale indicate a better outcome.
Change from baseline in parent rated view of their child's behavioral problems/defiant behavior | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent view of their child's behavioral problems/defiant behavior as measured by the Oppositional Defiant Scale of the Disruptive Disorder Rating Scale (DBD) which consists of 7 items rated on a 4-point scale ranging from 1 (not at all) to 4 (very much). Higher scores indicate a worse outcome.
Change from baseline in parent rated family warmth and conflict | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated warmth and conflict. Warmth and conflict are indexed by eight items rated on a five-point scale from 1 (never) to 5 (more than 7 times). Five items measure parent-child warmth and three items measure parent-child conflicts. Higher scores on parental warmth scale indicate a better outcome. Higher scores on the parent-child conflicts scale score indicate a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in parent rated encouragement of positive behaviors, setting limits, and proactive parenting behaviors | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated encouragement of positive behaviors, setting limits, and proactive parenting behaviors as indexed by the Parenting Children and Adolescents Scale (PARCA). The PARCA has 19 items rated on a five-point scale 1 = never to 5 = Very Often. The scale has three subscales on encouragement of positive behaviors, setting limits, and proactive parenting behaviors. Higher scores indicate a better outcome.
Change from baseline in parent rated stress | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated stress as measured by the Perceived Stress Scale (PSS). PSS consists of 10 questions about perceived stress during the last month rated on a 5-point Likert scale (0 = Never to 4 = Very Often). The scale measures the extent to which situations in one's life are assessed and perceived as stressful and current stress levels. Higher scores indicate a worse outcome.
Change from baseline in parent rated health | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated health as measured by the Hospital Anxiety and Depression Scale (HAD). HAD consists of two scales (a total of 14 items), one for anxiety and one for depression with seven questions each. Items are rated on a 4-point Likert scale. Higher scores indicate a worse outcome.
Change from baseline in parent rated parents validation of their child's emotions when expressed | Immediate PW group pretest in Fall 2022. Post test up to 10 months after pretest. Wait-list group pretest in Fall 2022. Post test 1 up to 10 months after pretest. Post test 2 for wait-list up to 10 months after post test 1
  Change from baseline up to 10 months later (immediate intervention group, two time points) and up to 20 months later (wait-list comparison group, three time points) in parent rated affective style as measured by the tolerating subscale of the Affective Style Questionnaire (ASQ). The ASQ consists of five items (rated on a 3 point Likert scale, 1 = Completely Agree to 3 = Completely Disagree) that examine how parents view their own validation of their child's emotions when expressed. Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ferrer-Wreder, PhD.,, Principal Investigator — Stockholm University
Locations (1):
- Stockholm University, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets to be collected in this trial are not readily available because this study's ethical review does not allow for study data to be in a public repository. For meta-analysis or confirmation of published study results, individual level, de-identified data requests will be reviewed when made by qualified researchers (e.g., Ph.D.) along with ethical permission under Swedish law regarding secondary data analysis. Requests to access the datasets should be directed to Laura Ferrer-Wreder (laura.ferrer-wreder@psychology.su.se)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will be made available after 6 months from the project completion date.
Access Criteria: The datasets to be collected in this trial are not readily available because this study's ethical review does not allow for study data to be in a public repository. For meta-analysis or confirmation of published study results, individual level, de-identified data requests will be reviewed when made by qualified researchers (e.g., Ph.D.) along with ethical permission under Swedish law regarding secondary data analysis. Requests to access the datasets should be directed to Laura Ferrer-Wreder (laura.ferrer-wreder@psychology.su.se)

REFERENCES:
- [Background] Goodman R. The Strengths and Difficulties Questionnaire: a research note. J Child Psychol Psychiatry. 1997 Jul;38(5):581-6. doi: 10.1111/j.1469-7610.1997.tb01545.x. PMID 9255702
- [Background] Malmberg M, Rydell AM, Smedje H. Validity of the Swedish version of the Strengths and Difficulties Questionnaire (SDQ-Swe). Nord J Psychiatry. 2003;57(5):357-63. doi: 10.1080/08039480310002697. PMID 14522609
- [Background] Pelham WE Jr, Gnagy EM, Greenslade KE, Milich R. Teacher ratings of DSM-III-R symptoms for the disruptive behavior disorders. J Am Acad Child Adolesc Psychiatry. 1992 Mar;31(2):210-8. doi: 10.1097/00004583-199203000-00006. PMID 1564021
- [Background] Criss MM, Shaw DS. Sibling relationships as contexts for delinquency training in low-income families. J Fam Psychol. 2005 Dec;19(4):592-600. doi: 10.1037/0893-3200.19.4.592. PMID 16402874
- [Background] Wetterborg D, Enebrink P, Lonn Rhodin K, Forster M, Risto E, Dahlstrom J, Forsberg K, Ghaderi A. A pilot randomized controlled trial of Internet-delivered parent training for parents of teenagers. J Fam Psychol. 2019 Oct;33(7):764-774. doi: 10.1037/fam0000541. Epub 2019 Jun 17. PMID 31204818
- [Background] Ringle JL, Mason WA, Oats RG, Cogua J. Parenting Children and Adolescents (PARCA) scale English to Spanish translation: An investigation of measurement invariance. J Fam Psychol. 2019 Dec;33(8):938-944. doi: 10.1037/fam0000559. Epub 2019 Jul 18. PMID 31318263
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Hofmann SG, Kashdan TB. The Affective Style Questionnaire: Development and Psychometric Properties. J Psychopathol Behav Assess. 2010 Jun 1;32(2):255-263. doi: 10.1007/s10862-009-9142-4. PMID 20495674
- [Derived] Olsson TM, Enebrink P, Kapetanovic S, Ferrer-Wreder L, Stalnacke J, Eninger L, Eichas K, Norman A, Lindberg L, Gull IC, Hau HG, Allodi MW, Sedem M. Study protocol for a non-randomized controlled trial of the effects of internet-based parent training as a booster to the preschool edition of PATHS(R): Universal edition of the Parent Web. PLoS One. 2023 Apr 27;18(4):e0284926. doi: 10.1371/journal.pone.0284926. eCollection 2023. PMID 37104280